CLINICAL TRIAL: NCT02047422
Title: A Prospective, Single-center, Randomized, Controlled, Open-label, Pilot Study to Compare the Effectiveness and Safety of DIuretics Add-On Strategy in Acute Decompensated Heart Failure Patients (DIOS II)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the diuretic which is planned to be used in the study is no longer available.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0808
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Congestive Heart Failure
Keywords: Heart failure, diuretics, kidney, glomerular filtration rate
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Metolazone; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Add furosemide/no spironolactone (Experimental)
  Interventions: Drug: Furosemide
- Add metolazone/no spironolactone (Experimental)
  Interventions: Drug: metolazone
- Add furosemid/spironolactone (Experimental)
  Interventions: Drug: furosemid/spironolactone
- Add metolazone/spironolactone (Experimental)
  Interventions: Drug: metolazone/spironolactone

INTERVENTIONS:
Drug: Furosemide — furosemide (doubling previous furosemide dose)
  Arms: Add furosemide/no spironolactone
Drug: metolazone — metolazone (add 2.5mg qod)
  Arms: Add metolazone/no spironolactone
Drug: furosemid/spironolactone — spironolactone (doubling previous spironoalctone dose or add 12.5mg BID if previous non-user)
  Arms: Add furosemid/spironolactone
Drug: metolazone/spironolactone — no spironolactone (maintaining previous spironolactone dose or not add spironolactone if previous non-user)
  Arms: Add metolazone/spironolactone

SUMMARY:
To compare the effectiveness and safety of diuretics add-on strategy in chronic heart failure patients

ELIGIBILITY:
Inclusion Criteria:

1. dyspnea at rest or minimal activity
2. tachypnea (respiratory rate > 20/min) or rales or pulmonary edema on chest X-ray

Exclusion Criteria:

1. hospitalization for acute heart failure decompensation
2. cardiogenic shock (Systolic Blood Pressure < 80mmHg)
3. Need or plan for renal replacement therapy (dialysis, kidney transplant)
4. serum creatine level > 2.5mg/dl
5. serum potassium (K+) > 5.5mg/dl
6. Age > 80 years old or poor compliance patients
7. allergy, adverse drug reaction, hypersensitivity to any kinds of diuretics
8. life expectancy < 6 months (e.g. metastatic malignancy, liver cirrhosis)
9. pregnancy or women at age of childbearing potential

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
urine output change | from admission to Hospital Day (HOD)#4
  efficacy of diuretics add-on therapy, urine output change

SECONDARY OUTCOMES:
serum creatinine change | from admission to HOD#4
  safety of diuretics add-on therapy, serum creatinine change

OTHER OUTCOMES:
body weight change | from admission to HOD#4
  body weight change, symptoms & signs change
urine creatinine change | from admission to HOD#4
  urine creatinine change, serum & urine electrolyte change, biomarkers change
clinical outcomes | at 90 days after discharge
  clinical outcomes ( all-cause mortality, all-cause rehospitalization, start of renal replacement therapy)